CLINICAL TRIAL: NCT05345054
Title: The Deep South Surgical Equity Research Network: Addressing Socioecological Determinants of Health
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Daniel Chu, Associate Professor, University of Alabama at Birmingham
Other Study IDs: 300009121
Record Dates: First submitted 2022-04-02; First posted 2022-04-25 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer; Inflammatory Bowel Diseases; Diverticular Diseases; Social Behavior
MeSH Terms: conditions — Colorectal Neoplasms; Inflammatory Bowel Diseases; Diverticular Diseases; Social Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Phase 1: Study Population and Enrollment. To ensure survey feasibility and acceptability for our target population we will purposively recruit older African American patients at each of the three participating sites. Using conservative estimates of clinical volume as well as US county level census data we estimate enrolling 3 elderly (>65 years of age) African American participants per site per week with a target enrollment of 12 patients per site.
  Interventions: Other: no intervention
- Phase 2: To gain a broad understanding of barriers to surgical access and care in the Deep South, each study site will conduct key informant interviews. Participants will be recruited from five socioecological levels: patient, caregivers/provider, organizational, community, and policy-levels. At each site, two key informant interviews will be performed at each socioecological level (2 patients, 2 caregivers, 2 providers, 2 organizational leaders, 2 community leaders, and 2 policy leaders = 12 per site). We will purposively sample 100% of the participants at the patient and caregiver level (n=12) to be African American and >65 years old.
  Interventions: Other: no intervention
- Phase 3: Enrollment Process. Eligibility criteria for this phase of study enrollment will be broadened to include all English-speaking patients >18 years of age undergoing or having recently undergone (<7 days) an ACS-NSQIP defined surgical procedure. At each site, eligible participants will be approached by a trained research associate pre-operatively in clinic (for elective cases) or post-operatively in the hospital (for emergency cases <7 days). Because each enrollment site has a unique schedule, site representatives will coordinate the most efficient weekly schedule.
  We expect to reach our target enrollment (100 participants total, 33 at each site) in 1 year based on conservative estimates of clinical case volume. We expect to enroll at least 20% elderly participants (>65 years of age) and between 30-50% African American participants based on county level (Greenville - Butler County, Demopolis - Marengo County, Alexander City - Tallapoosa County) census data.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — This study will not involve an intervention of any sort. Participants will either take a survey or undergo an interview, and those taking the survey will have clinical data captured.
  Other Names: no intervention planned

SUMMARY:
Rationale: Older African Americans undergoing surgery are a vulnerable and growing population at high risk for poor surgical outcomes and disparities. Few programs have focused on this population due to a fragmented understanding of the needs of this population.

Objectives: While socioecological determinants of health (SEDOH) such as health literacy and socioeconomic status are known drivers of surgical disparities, an estimated 36-47% of surgical disparities remains unexplained. This gap results from limitations of current clinical datasets in capturing SEDOHs. This pilot study aims to fill this gap by (i) collecting granular SEDOH data, (ii) identifying barriers to surgical care for older African Americans, and (iii) establishing a multi-institutional clinical database through a socioecological context. These findings will help understand how SEDOHs drive surgical disparities and inform development of interventions to eliminate them in elderly African Americans.

Design and Methods: Guided by the socioecological model of health, the investigators will use mixed-methods to achieve the objectives. First, the investigators will assess the acceptability and feasibility of a 58-item SEDOH survey based on the NIH PhenX toolkit. After distributing this survey to 36 elderly (≥65 years) African American patients undergoing surgery at 3 rural, UAB-affiliated hospitals (Alex-City, Greenville, Demopolis) the investigators will conduct detailed theory guided assessments of acceptability and feasibility (SA1). Second, the investigators will conduct key informant interviews of individuals from all 5 socioecological levels at each rural hospital (n=10) to identify additional barriers and facilitators to surgical care. The investigators will purposively sample 100% of participants at the patient and caregiver level (n=12) to be elderly African Americans (SA2). Finally, the investigators will link measured SEDOH data with standardized clinical data at each hospital to establish a novel database (SA3). These findings will establish a process to measure SEDOHs across the Deep South and set the foundation for a unique database to study surgical disparities.

Significance: Development of effective multilevel interventions to eliminate surgical disparities in older African Americans is dependent on a clearer understanding of the contextual drivers of these disparities. This pilot study will accelerate understanding of these mechanism(s) through SEDOHs. It will establish a process to measure SEDOHs, identify additional barriers to surgical care not captured by NIH instruments, and build the database to study these relationships. Such findings will have the potential to impact vulnerable surgical populations in the Deep South and support the Deep South RCMAR mission to promote health and optimize health outcomes for older and rural African Americans.

ELIGIBILITY:
Inclusion Criteria for Patients for Phase 1 and 2

-≥ 65 years old undergoing or having recently undergone colorectal surgery* (<7 days) for colorectal disease**

* All genders
* African American race
* Able to consent
* English-speaking

Exclusion Criteria for Patients for Phase 1 and 2

* <65 years old
* Race other than African American
* Undergoing operation other than colorectal surgery
* Unable to consent
* Limited mental state

Inclusion Criteria for other participants in Phase 2

-≥ 18 years old

* All genders
* All race/ethnicities
* Able to consent English-speaking

Exclusion Criteria for other participants in Phase 2

* Child (<18 years)
* Unable to consent
* Limited mental state

Inclusion Criteria for Phase 3

* ≥ 18 years old undergoing or having recently undergone colorectal surgery* (<7 days) for colorectal disease**
* All genders
* All race/ethnicities
* Able to consent
* English-speaking

Exclusion Criteria for Phase 3

* Child (<18 years)
* Undergoing operation other than colorectal surgery
* Unable to consent
* Limited mental state

  * Includes colectomy/proctectomies. ** Includes colorectal cancer, inflammatory bowel disease and diverticular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients for participation in Phases 1, 2, and 3 will be selected from those undergoing colorectal surgery at UAB affiliated sites in Alabama (Demopolis, Greenville, Alexander City).
  Additional participants for Phase 2 will come from all other socioecological levels (caregiver, provider, organizational leaders, community leaders, public policy/governmental leaders).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-08-12 (Actual)

PRIMARY OUTCOMES:
Feasibility and Acceptability of a multidimensional survey in measuring socioecological determinants of health at rural hospitals in the Black Belt of Alabama (Demopolis, Alexander City, Greenville). | 3 months
  Using a theory guided framework and previously published measures of acceptability and feasibility, a post survey will be administered to all participants in specific aim 1. Feasibility and acceptability scores will be calculated, with positive acceptability and feasibility being indicated by scores of 4 or greater on a likert scale. The investigators will ensure that the survey is found to be acceptable and feasible to >70% of the target population, and will have areas for qualitative feedback and comments to adapt the survey as needed.
Barriers to surgical care for older African American patients in the Deep South. | 6 months
  To identify barriers to surgical care for older African American patients in the Deep South the investigators will conduct qualitative interviews of participants at all socioecological levels at each site. These interviews will be transcribed and coded using NVivo software, and themes from this analysis will be compared with the domains assessed in the survey used in specific aim 1 in order to ensure that all relevant domains are captured and assessed.
A database linking socioecological determinants of health with nationally validated surgical outcomes. | 12 months
  To establish a database linking socioecological determinants of health with nationally validated surgical outcomes the investigators will pair data obtained from the previously developed survey with chart abstracted clinical outcomes data. All data will be stored in a secure RedCap database, and entered only by trained abstractors.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Chu, MD, Principal Investigator — University of Alabama in Birmingham
Locations (3):
- United States (3):
  - Russell Medical Center, Alexander City, Alabama
  - Whitfield Regional Medical Center, Demopolis, Alabama
  - Regional Medical Center of Central Alabama, Greenville, Alabama

IPD SHARING:
Plan to Share IPD: No
Primary data acquired through the quantitative surveys and other demographics will be collected and managed using REDCap (Research Electronic Data Capture). As the host/coordinating center, UAB REDCap servers are secured through a virtualized environment behind an enterprise grade Palo Alto firewall. Only IRB-approved research team members will have access to the REDCap system through a secure and unique login. UAB REDCap is in compliance with NIST 800-53/800-171 (HIPAA) and FDA CFR21 part 11 guidelines, approved by all authorizing parties at UAB and authorized to operate (ATO) from NIH/NHLBI.